CLINICAL TRIAL: NCT04836351
Title: Feasibility, Usefulness and Evaluation of a Concentrated Rehabilitation for Patients With Persistent Symptoms Post COVID-19
Brief Title: Rehabilitation for Patients With Persistent Symptoms Post COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western Norway University of Applied Sciences (Other)
Collaborators: Helse-Bergen HF (Other)
Responsible Party: Principal Investigator, Kiri Lovise Njøten, Ph.d student, Western Norway University of Applied Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WesternNorwayUAS
Record Dates: First submitted 2021-03-29; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Covid19
Keywords: long COVID; post-acute COVID syndrome; persistent symptoms post COVID-19
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: Feasibility study, one group pre-post design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Concentrated rehabilitation (Experimental): 3+ 1-2 day concentrated rehabilitation for patients with persistent symptoms post COVID-19.
  Interventions: Other: Concentrated rehabilitation for patients with persistent symptoms post COVID-19

INTERVENTIONS:
Other: Concentrated rehabilitation for patients with persistent symptoms post COVID-19 — 3+ 1-2 days concentrated rehabilitation for patients with persistent symptoms post COVID-19 with a mobile application follow-up and physical consultations at 3 months post intervention.

SUMMARY:
A large proportion of persons who have had COVID-19 have reported persisted symptoms as fatigue and dyspnea months post infection which affect activities of daily living.

The aim of the study is to examine the feasibility and safety of a concentrated rehabilitation program with a mobile application follow-up for persons with persistent symptoms post COVID-19 infection. We will examine recruitment availability, adherence to the program, goal achievement, and resources requirements.

Methods: A feasibility study with one group pre-post test design with 10-20 persons between 18-67 years, with persistent symptoms post COVID-19 will be included. The intervention is 3+ 1-2 days concentrated rehabilitation with a mobile application follow-up for 3 months.

Following assessments wil be used: Cardiopulmonary exercise testing, lung function, functional performance tests, questionnaires regarding dyspnea, fatigue, anxiety, depression, work-status, health status, sleep behavior, physical activity level.

Demographic data before and after the intervention will be presented. Focus group interview will be done with the participants. The interview will be analysed using systematic text condensation.

DETAILED DESCRIPTION:
In March 2020, the World Health Organization (WHO) declared the COVID-19 outbreak to be a pandemic, and a year later more than 120 000 000 people are confirmed with the disease. The disease has caused more than 2 700 000 deaths globally. Norway has a low mortality rate compared to rest of the world. However, a large proportion (10-33%) of the patients worldwide have reported persistent symptoms, such as dyspnea, reduced exercise capacity, loss of taste/smell and fatigue months after the infection. Persistent symptoms are also found in younger populations and in persons with an initially mild disease.

The intervention will take place at "Helse i Hardanger" (HiH)(Health center in Hardanger, Norway). The participants will stay for a 3 -day rehabilitation intervention, if needed, another 1 or 2-day stay will be offered about a month later. The concentrated treatment will be given by an interdisciplinary team, including doctors, physiotherapists, nutritionists, pharmacists, psychologists/psychiatrists, and nurses. The intervention is an individualized group treatment based on behavioural change.

ELIGIBILITY:
Inclusion Criteria:

* persistent symptoms minimum 2 months post COVID-19 infection
* reduced exercise capacity level
* symptoms of dyspnea and/or fatigue

Exclusion Criteria:

* diseases where exercise is contraindicated (e.g. unstable angina pectoris)
* drug abuse, severe mental illness where treatment in groups are contraindicated.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary exercise test (CPET) | 4 months
  CPET performed at treadmill
Chalder Fatigue Questionnaire (CFQ) | 4 months
  Assessing fatigue

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | 4 months
  Assessing physical activity
Generalized Anxiety Disorder (GAD-7) | 4 months
  Evaluation of mental disorders
Patient Health Questionnaire (PHQ-9) | 4 months
  Assessing health status
Bergen Insomnia Scale (BIS) | 4 months
  Assessing sleep behavior
Client Satisfaction Questionnaire (CSQ-8) | 3 months
  Assessing client satisfaction with the treatment
Work and Social Adjustment Scale (WSAS) | 4 months
  Assessing ability to work and leisure activities.
The Brief Illness Perception Questionnaire (BIPQ) | 4 months
  Assessing the cognitive and emotional representations of illness.
Modified Medical Research Council Dyspnea Scale (mMRC) | 4 months
  Assessing dyspnea
Dyspnea-12 | 4 months
  Assessing dyspnea
Stair Climbing Test (SCT) | 4 months
  Evaluation of functional exercise capacity
30 second sit to stand test (30STST) | 4 months
  Evaluation of functional exercise capacity
Spirometry, plethysmography and maximal voluntary ventilation | 4 months
  Evaluation of lung function
Bioimpedance measurement | 4 months
  Assessment of body composition

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Kvale, PhD, Study Chair — University of Bergen
Locations (1):
- Helse i Hardanger, Øystese, Kvam Herad, Norway

IPD SHARING:
Plan to Share IPD: No
In accordance with the approvals granted for this study by The Regional Committee on Medical Research Ethics and The Norwegian Data Inspectorate, the data files are stored securely and in accordance with the Norwegian Law of Privacy Protection. A subset of the data file with anonymized data can be made available to interested researchers upon reasonable request to Bente Frisk providing Norwegian privacy legislation and General Data Protection Regulation (GDPR) are respected, and that permission is granted from The Norwegian Data Inspectorate and the data protection officer Western Norway University og Applied Sciences